CLINICAL TRIAL: NCT07339332
Title: A Clinical Study Exploring the Safety, Efficacy and Cell Metabolic Dynamics of Universal CD19 / 20 Car-t Cell Injection in Moderate to Severe Refractory Systemic Lupus Erythematosus
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Qiubai Li, Director, Head of Department of Rheumatology and Immunology, Principal Investigator, Professor, Wuhan Union Hospital, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT1195E-CG11009
Record Dates: First submitted 2025-11-18; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT1195E CAR-T cells Injection (Experimental): CT1195E cells infusion
  Interventions: Other: CAR-T Therapy

INTERVENTIONS:
Other: CAR-T Therapy — CT1195E cells infusion

SUMMARY:
This study is a single arm, open, exploratory dose escalation clinical study to evaluate the safety, efficacy, and cellular metabolic dynamics of ct1195e cells in patients with SLE.

DETAILED DESCRIPTION:
The study was divided into dose increasing stage and dose expanding stage.dose escalation phaseThree dose levels are tentatively determined for dose escalation: 3.0 × 108, 4.5 × 108 and 6.0 × 108 car-cd19/CD20+T cells. It is estimated that the target toxicity probability of the maximum tolerated dose is 30%, and about 12 participants are planned to be enrolled, and the number of enrolled patients in each dose group is subject to the actual situation. During the test, the researchers and partners will jointly negotiate whether to increase or decrease the dose, whether to increase to the set maximum dose group or produce the maximum available cell volume, and whether to increase the exploration of new dose level within the explored dose range (allowed to be conducted when the dose is increased or decreased) according to the participants' cell metabolism characteristics, safety, tolerance and preliminary effectiveness data, so as to determine the possible recommended therapeutic dose (RD).The DLT observation period is 28 days after the first infusion. If the treatment needs to be withdrawn before 28 days after the infusion due to disease progression or other reasons, no obvious car-t cell expansion is detected or car-t treatment is invalid, and the DLT related AE events determined by the researcher may not be related to the product, the DLT observation period can be completed before. During each dose increase, if there is a safety risk that needs to be discussed, the researchers and partners can make a dose increase/stability/decrease decision according to the safety and tolerance of participants and the metabolic kinetics of ct1192 cells. In the same dose group, the first participant had no significant safety risk 14 days after the completion of cell infusion, and subsequent participants could only carry out cell infusion.dose expansion phaseOne or more dose groups may be selected for dose expansion according to the results of the dose increasing stage to further explore the efficacy and safety in SLE patients. Each dose group and each queue plan to include up to 9 cases, and the specific number of patients in the group is subject to the actual number. DLT will not be observed in the dose expansion phase, and other research processes are the same as the dose increment phase. Researchers and collaborators will continue to monitor the safety data of the whole dose expansion phase and make decisions on admission and exit when necessary.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signing of Informed Consent Form (ICF): I fully understand and am informed of this study, and I have signed the Informed Consent Form, expressing my willingness to follow and complete all research procedures;
* When signing the ICF, the age should be between 18 and 65 years old (inclusive), with no gender restrictions;
* No systemic active infection (such as infectious pneumonia, tuberculosis) within 2 weeks before screening;
* Females with fertility (defined as all females who are physiologically capable of becoming pregnant) must agree to use highly effective contraception from at least 28 days before the start of self-cleaning to 1 year after CT1195E infusion, and absolutely prohibit egg donation within 1 year after receiving study treatment during the study period. Their male partners with fertility must agree to use effective barrier contraception from the start of self-cleaning to 1 year after CT1195E infusion, and should not donate semen or sperm during the entire study period;
* Females with fertility must have a negative serum beta-human chorionic gonadotropin (β-hCG) test result at screening and within 48 hours prior to the initiation of chemotherapy.
* Meet the EULAR/ACR 2019 classification criteria for SLE, with a disease history of ≥6 months;
* Prior to screening, patients must have received treatment with glucocorticoids combined with immunosuppressants (including cyclophosphamide, mycophenolate mofetil, tacrolimus, methotrexate, cyclosporine, leflunomide) and/or biologics for ≥3 months, with a stable dosage for ≥2 weeks, and the disease must still be in an active state. During screening, oral steroids must meet the following requirements:

If treated with hormone therapy alone, prednisone (or equivalent medication) should be ≥7.5 mg/day; When used in combination with immunosuppressants and/or biologics, there is no minimum daily dosage requirement for steroids;

* During screening, positive for antinuclear antibody, and/or positive for anti-ds-DNA antibody, and/or positive for anti-Smith antibody;
* During the screening period, patients with a SLEDAI-2K score of ≥7, or those with concurrent significant organ dysfunction, such as severe immune-mediated thrombocytopenia, lupus nephritis (histologically diagnosed as active nephritis type III or IV with or without type V);
* During screening, involvement of active organs (including kidneys, heart and lungs, musculoskeletal system, blood system, blood vessels, etc.; involvement of skin and mucous membranes alone is not included) is present;
* Adequate organ function:

  1. Renal function: defined as creatinine clearance rate (Cockcroft-Gault) calculated without hydration assistance ≥ 50 mL/min;
  2. Bone marrow function: defined as absolute neutrophil count (ANC) ≥1.0×10^9/L and hemoglobin (Hb) ≥60 g/L. During the 7 days prior to screening for inclusion and exclusion criteria, blood transfusions and growth factors must not be used to meet these requirements;
  3. Liver function: defined as alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels ≤2× upper limit of normal (ULN), and total bilirubin levels ≤2× upper limit of normal (ULN)
  4. Coagulation function: defined as an international normalized ratio (INR) or activated partial thromboplastin time (APTT) ≤1.5×ULN;
  5. Lung function: When exposed to indoor air, the blood oxygen saturation (SpO2) is ≥92% (measured by a pulse oximeter);
  6. Cardiac function: defined as having a left ventricular ejection fraction (LVEF) of ≥50% as assessed by echocardiography (ECHO) within the 8 weeks prior to screening.

Exclusion Criteria:

* Those who have suffered from severe lupus nephritis within the previous 2 months and require hemodialysis, or have received prednisone ≥100 mg/d or equivalent hormone treatment for ≥14 days;
* Those who have undergone plasma exchange, plasma separation, hemodialysis within the previous 30 days, or those who have suffered from lupus crisis within the previous 30 days;
* Screen for individuals with a history of ≥ Grade 2 bleeding within the previous 30 days or those requiring long-term anticoagulant therapy;
* History of any of the following cardiovascular diseases within 30 days prior to screening: heart failure of NYHA class III or IV, myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmias, any ventricular arrhythmias, or other clinically significant heart diseases;
* Before screening, there were manifestations of the central nervous system caused by lupus, including but not limited to lupus headache, seizures, cognitive impairment, impaired intellectual function, and visual impairment;
* Individuals with central nervous system diseases prior to screening include, but are not limited to: cerebrovascular accident, encephalitis, epilepsy, convulsion/seizure, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, central nervous system vasculitis, cognitive dysfunction, brain organic syndrome, or psychosis;
* Screen for the absence of systemic active infections within the previous 2 weeks, including but not limited to active tuberculosis;
* Previous exposure to CAR-T cell therapy or other gene-modified T cell therapies, or a history of major organ transplantation (such as heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation;
* Allergic or intolerant to diuretics, tocilizumab, or experiencing life-threatening allergic reactions, hypersensitivity reactions, or intolerance to CT1195E formulation or its excipients (including dimethyl sulfoxide (DMSO)), or having a history of other severe allergies such as anaphylactic shock;
* Screen for individuals who have used targeted B-cell drugs such as rituximab within the previous 3 months;
* Exclusion criteria: Subjects who have used other biologics such as TACI-Ig and Benlysta within the previous 12 weeks;
* Within 2 weeks prior to the infusion of CT1195E, the use of prednisone (or equivalent drugs) at a dosage of ≥10 mg/day is allowed. Physiological substitutes, topical, and inhaled steroids are also permitted;
* Received T-cell-affecting immunosuppressants (mycophenolate mofetil, methotrexate, cyclosporine, azathioprine, leflunomide, tacrolimus) within 2 weeks before infusion of CT1195E;
* Have received JAK inhibitors (such as tofacitinib, baricitinib, ruxolitinib, etc.) within 2 weeks before the infusion of CT1195E;
* Have received attenuated live vaccine, inactivated vaccine, or RNA vaccine within one month before screening;
* Suffered from malignant tumor within 2 years before signing the ICF. The following conditions are excluded: non-melanoma skin cancer that has undergone radical treatment, localized prostate cancer, biopsy-confirmed cervical carcinoma in situ or squamous intraepithelial lesion detected by cervical smear, and completely resected breast carcinoma in situ;
* The participant has undergone major surgery within 4 weeks prior to signing the informed consent form, or plans to undergo major surgery during the study period, and the investigator believes that this would pose an unacceptable risk to the study participant;
* During screening, there is evidence of HIV, syphilis infection, active hepatitis B virus infection (HBsAg positive and HBV-DNA above the detection limit), or active hepatitis C virus infection (both HCV antibody and HCV-RNA positive);
* Those who participated in other clinical studies within the previous three months or are still within the five half-lives after the last dose;
* Concurrent major chronic diseases that are not under control and that the investigator believes may increase the risk to study participants;
* Subjects with a history or evidence of suicidal thoughts within the previous 6 months, or any suicidal behavior within the previous 12 months, are considered by the researchers to have a significant risk of suicide;
* Pregnant or lactating women;
* The researcher judges that the study participant has poor compliance, is unable or unwilling to adhere to the requirements of the study protocol, or has other reasons that make them unsuitable for participating in this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
severity of dose limiting toxicity (DLT) | Within 28 days after infusion
Incidence of dose limiting toxicity (DLT) | Within 28 days after infusion
Evaluate the maximum tolerable dose (MTD) and/or dose range of ct1195E | After medication to day 28
  Ct1195E MTD and/or dose range
severity of adverse events (AES) | Within 180 days after infusion
Incidence of adverse events (AES) | Within 180 days after infusion

SECONDARY OUTCOMES:
Proportion of participants with SLE responder index (sri-4) | 1, 2,3, 6, 9 and 12 months after drug use
  Preliminary evaluation of the efficacy of ct1195E in the treatment of moderate to severe refractory SLE.Proportion of participants who reached SLE responder index (sri-4) at 6 months and other time points (1, 2,3, 9 and 12 months after medication)
Proportion of participants with low lupus disease activity status (lldas) | 1, 2,3, 6, 9 and 12 months after drug use
  To evaluate the efficacy of ct1195E in the treatment of moderate to severe refractory SLE. The proportion of participants who reached lupus low disease activity status (lldas) at 6 months and other time points (1, 2, 3, 9 and 12 months after medication).
Proportion of participants achieving disease remission (doris) | 1, 2, 3, 6, 9 and 12 months after drug use
  To evaluate the efficacy of ct1195E in the treatment of moderate to severe refractory SLE. The proportion of participants who achieved disease remission (doris) at 6 months and other time points ((1, 2, 3, 9 and 12 months after medication).
Changes of SLE disease activity index (sledai-2k) score from baseline after medication | 1,2,3,6,9 and 12 months after drug use
  The score range of the Health Assessment Questionnaire Disability Index (HAQ-DI) is usually 0 to 3, where 0 represents no disability or intact function, and 3 represents severe disability or complete loss of function. The higher the score, the worse the functional status of the patient, that is, the higher the degree of disability; Conversely, the lower the score, the better the function.
After treatment, the SLE disease activity index (Selena - SLEDAI) score changed from baseline | 1, 2, 3, 6, 9 and 12 months after drug use
  The minimum value of selena-sledai score is 0 points, and the maximum value can reach 105 points theoretically, but in actual clinical practice, 10 to 15 points usually indicate the presence of disease activity. Higher scores indicate higher disease activity rather than better outcomes. The score is used to quantify the activity of systemic lupus erythematosus (SLE). An increase in the score reflects a more active condition, which requires active clinical intervention; Conversely, a reduced score indicates good disease control.
After treatment, the index of lupus erythematosus assessment group (bilag-2004) changed from baseline | 1, 2, 3, 9 and 12 months after drug use
  The minimum value of the British Isle lupus rating group index (bilag-2004) is 0 and the maximum value is 100. The higher the score, the higher the disease activity, that is, the more serious the disease.
The SLE activity score (sle-das) changed from baseline after treatment | 1, 2, 3, 9 and 12 months after drug use
  The minimum value of sle-das score (systemic lupus erythematosus disease activity score) is 0, and the maximum value is usually 100. This score quantifies the disease activity by accumulating the scores of clinical and laboratory indicators. The higher the score, the stronger the disease activity and the more serious the disease.
Changes in clinicians' overall judgment (PGA) score from baseline after medication | 1, 2, 3, 9 and 12 months after drug use
  In systemic lupus erythematosus (SLE), the minimum value of the doctors' global assessment (PGA) score is 0, and the maximum value is 3, where 0 indicates no disease activity and 3 indicates the most serious disease activity. The higher the score, the higher the disease activity, that is, the worse the result; Conversely, the lower the score, the lower the disease activity, and the better the result.
Proportion of patients without other SLE therapy after medication | 1, 2, 3, 9 and 12 months after drug use
Changes in immunoglobulin (IgG, IgM, IgA) levels during medication | 1, 2, 3, 9 and 12 months after drug use
The change value of post medication Health Assessment Questionnaire Disability Index (HAQ-DI) from baseline | 1, 2, 3, 9 and 12 months after drug use
  The minimum possible score of patients with systemic lupus erythematosus (SLE) using the Health Assessment Questionnaire Disability Index (HAQ-DI) is 0, and the maximum possible score is 3; The higher the score, the more severe the dysfunction of the patient, that is, the worse the outcome.
duration of ct1195E gene in blood | Within 1 year after CAR-T cell infusion
  Objective to evaluate the cell kinetics of ct1195E in SLE participants, and to observe the level and duration of ct1195E gene copy number in blood.
Copy numbe of ct1195E gene in blood | Within 1 year after CAR-T cell infusion
  Objective to evaluate the cell kinetics of ct1195E in SLE participants, and to observe the level and duration of ct1195E gene copy number in blood.
Changes of B cell functional subsets (initial B cells, memory B cells, plasma cells) after ct1195E infusion | Within 1 year after CAR-T cell infusion
  Evaluate the efficacy (PD) characteristics of CT1195E in SLE participants. Changes in the levels of B cell functional subgroups (initial B cells, memory B cells, plasma cells) after CT1195E infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospita, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No